CLINICAL TRIAL: NCT00347477
Title: Fluid Shift in Patients Treated With Therapeutic Hypothermia After Cardiac Arrest, and How do They Manage Life Afterwards?
Brief Title: Fluid Shifts in Patients Treated With Therapeutic Hypothermia After Cardiac Arrest
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Bård E Heradstveit, MD, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12080
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-03

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; hypothermia; neurologic outcome; edema
MeSH Terms: conditions — Heart Arrest; Hypothermia; Edema

INTERVENTIONS:
Drug: HyperHAES vs. RA-solution/NaCl

SUMMARY:
Therapeutic hypothermia after cardiac arrest har shown to improve the rate of survival in a significant way. However hypothermia also causes leak of fluid into the surrounding tissue. This edema could lead to damage to the same tissue, not beneficial for the patients. We therefore try to evaluate if hyperosmolar, hyperoncotic fluid as an alternative to std. treatment (NaCl/RA)could affect the edema in a positive way, and result to a better outcome neurological for the patients.

DETAILED DESCRIPTION:
After the patients are admitted to our hospital we randomise them to either std. fluid therapy (NaCl/RA) or HyperHAES. After PCI we state the rate of cerebral edema by carrying out a cerebral MRI before the cooling starts. We treat the patients with the different fluids for 24 hours. We then evaluate the edema after 24 and 72 hours by the same method. In addition we state the rate of peripheral capillary leak by Wick'S method. The capillary leak is calculated every 8.th hour for the 1. day the patients are treated in our ICU. AFter 1 year, those who survive are invited to a follow-up where we test the patient using Mini MEntal Status, SF-36, in addition to neurophysiological tests as EEG and the P300-test. We then relate the results to the fluid given initially after the cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed cardiac arrest,
* ALS started within 15 min.
* ROSC within 60 min.
* Still unconscious,
* Age 18-80

Exclusion Criteria:

* Other malignancies,
* Persons who wake up,
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-04 (Actual); Study Completion 2009-03

PRIMARY OUTCOMES:
Mortality
Quality of Life

SECONDARY OUTCOMES:
Days in the ICU
Neurological test as described
Grade of Edema

CONTACTS AND LOCATIONS:
Overall Officials: Jon k Heltne, Dr.med, Study Chair — AKuttmedisin/KSK/ Haukeland University Hosp.
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Heradstveit BE, Guttormsen AB, Langorgen J, Hammersborg SM, Wentzel-Larsen T, Fanebust R, Larsson EM, Heltne JK. Capillary leakage in post-cardiac arrest survivors during therapeutic hypothermia - a prospective, randomised study. Scand J Trauma Resusc Emerg Med. 2010 May 25;18:29. doi: 10.1186/1757-7241-18-29. PMID 20500876